CLINICAL TRIAL: NCT06430606
Title: How Do Novel Oxygenation Indices Change with Trendelenburg Position in Robot-Assisted Laparoscopic Surgeries?
Brief Title: Novel Oxygenation Indices in Robot-Assisted Laparoscopic Surgeries
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Furkan Tontu, Doctor of Anesthesiology and Reanimation, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-05-
Record Dates: First submitted 2024-05-15; First posted 2024-05-28 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Ventilator-Induced Lung Injury
Keywords: trendelenburg; robot-assisted laparoscopic surgery
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing robotic-assisted laparoscopic surgery: The patients consist of ASA I-II or III group undergoing robotic-assisted laparoscopic surgery.
  Interventions: Procedure: Tint Time; Procedure: T0 Time; Procedure: T1

INTERVENTIONS:
Procedure: Tint Time — Arterial blood gas was obtained immediately after intubation(Tint) in supine position. Ventilator parameters and hemodynamic parameters were recorded.
Procedure: T0 Time — Arterial blood gas was obtained immediately after pneumoperitoneum in trendelenburg position. Ventilator parameters and hemodynamic parameters were recorded.
Procedure: T1 — Arterial blood gas was obtained immediately after pneumoperitoneum in trendelenburg position. Ventilator parameters and hemodynamic parameters were recorded.

SUMMARY:
In this study, changes in new oxygenation indices investigated by Asar et al. will be compared with conventional oxygenation and saturation indices in patients undergoing robot-assisted laparoscopic surgery due to pneumoperitoneum and Trendelenburg position.

DETAILED DESCRIPTION:
During the intraoperative period, optimal oxygenation should be achieved while avoiding the harmful effects of hypoxia and hyperoxia in patients. The PaO2/FiO2 and SpO2/FiO2 ratios have been traditionally used to assess this condition. Subsequently, oxygenation indices incorporating mean airway pressure have been developed, such as the oxygenation index (OI = (FiO2 × Pmean) / PaO2) and oxygenation saturation index (OSI = (FiO2 × Pmean) / SpO2). More recently, Asar et al. have defined 8 novel oxygenation indices using mean power (MP) and driving pressure (DP) instead of Pmean (OSI-MPtot, OI-MPtot, OSI-ΔPinsp, OI-ΔPinsp, OSI-MPdyn, OI-MPdyn, PaO2/(FiO2xPEEP), and SpO2/FiO2xPEEP). They compared the predictive power of these new indices for intensive care unit (ICU) mortality in COVID-ARDS (C-ARDS) patients with conventional oxygenation indices (PaO2/FiO2, SpO2/FiO2, OI, OSI). OI-ΔPinsp, OSI-ΔPinsp, and OSI-MPdyn indices were found to have the highest predictive power for ICU mortality. However, there is currently no study investigating the changes of these new indices during the intraoperative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class I-III
* Age between 18-75 years
* Signed informed consent form

Exclusion Criteria:

* Diagnosis of COPD (Chronic Obstructive Pulmonary Disease) and asthma
* History of thoracic surgery
* Body mass index (BMI) > 35
* Development of hemodynamic instability or desaturation (SpO2 < 92) during the operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population The study will include 42 volunteer patients, aged over 18, classified under the American Society of Anesthesiologists Physical Status Classification (ASA) I-III risk groups, who are scheduled to undergo robot-assisted laparoscopic surgery at the Health Sciences University Basaksehir Cam and Sakura City Hospital operating room.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum OSI-MPtot in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OI-MPtot in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OSI-ΔPinsp in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OI-ΔPinsp in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OSI-MPdyn in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OI-MPdyn in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on PaO2/(FiO2xPEEP) in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on SpO2/FiO2xPEEP in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on SpO2/FiO2 in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OI (oxygenation index) in ASA I-III patients undergoing robot-assisted laparoscopic surgery.
Oxygenation indices | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  This study aims to investigate the effects of Trendelenburg position and pneumoperitoneum on OSI (oxygenation saturation index) in ASA I-III patients undergoing robot-assisted laparoscopic surgery.

SECONDARY OUTCOMES:
Mechanical ventilator parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in PEEP (cmH2O) with Trendelenburg position and pneumoperitoneum
Mechanical ventilator parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in compliance (mL/cmH2O) with Trendelenburg position and pneumoperitoneum
Mechanical ventilator parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in peak pressure (cmH2O) with Trendelenburg position and pneumoperitoneum
Arterial blood gas parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the pH with Trendelenburg position and pneumoperitoneum
Arterial blood gas parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the base excess(mmol/lt) with Trendelenburg position and pneumoperitoneum
Arterial blood gas parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the partial oxgyen(mmHg) with Trendelenburg position and pneumoperitoneum
Arterial blood gas parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the partial carbon dioxide(mmHg) with Trendelenburg position and pneumoperitoneum
Arterial blood gas parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the lactate(mmol/lt) with Trendelenburg position and pneumoperitoneum
Hemodynamic parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the heart rate with Trendelenburg position and pneumoperitoneum
Hemodynamic parameters | during the surgery and immediately after the surgery (approximately 3 hours to 6 hours)
  Change in the mean arterial blood pressure with Trendelenburg position and pneumoperitoneum

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Background] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583
- [Background] Queiroz VNF, da Costa LGV, Barbosa RP, Takaoka F, De Baerdemaeker L, Cesar DS, D'Orto UC, Galdi JR, Gottumukkala V, Cata JP, Hemmes SNT, Hollman MW, Kalmar A, Moura LAB, Mariano RM, Matot I, Mazzinari G, Mills GH, Posso IP, Teruya A, Vidal Melo MF, Sprung J, Weingarten TN, Treschan TA, Koopman S, Eidelman L, Chen LL, Lee JW, Arino Irujo JJ, Tena B, Groeben H, Pelosi P, de Abreu MG, Schultz MJ, Serpa Neto A; AVATaR and PROVE Network investigators. International multicenter observational study on assessment of ventilatory management during general anaesthesia for robotic surgery and its effects on postoperative pulmonary complication (AVATaR): study protocol and statistical analysis plan. BMJ Open. 2018 Aug 23;8(8):e021643. doi: 10.1136/bmjopen-2018-021643. PMID 30139899
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Biehl M, Binnekade JM, Canet J, Fernandez-Bustamante A, Futier E, Gajic O, Hedenstierna G, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Putensen C, Ranieri M, Scavonetto F, Schilling T, Schmid W, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network Investigators. Protective versus Conventional Ventilation for Surgery: A Systematic Review and Individual Patient Data Meta-analysis. Anesthesiology. 2015 Jul;123(1):66-78. doi: 10.1097/ALN.0000000000000706. PMID 25978326
- [Background] O'Gara B, Talmor D. Perioperative lung protective ventilation. BMJ. 2018 Sep 10;362:k3030. doi: 10.1136/bmj.k3030. PMID 30201797
- [Background] Tartler TM, Ahrens E, Munoz-Acuna R, Azizi BA, Chen G, Suleiman A, Wachtendorf LJ, Costa ELV, Talmor DS, Amato MBP, Baedorf-Kassis EN, Schaefer MS. High Mechanical Power and Driving Pressures are Associated With Postoperative Respiratory Failure Independent From Patients' Respiratory System Mechanics. Crit Care Med. 2024 Jan 1;52(1):68-79. doi: 10.1097/CCM.0000000000006038. Epub 2023 Sep 11. PMID 37695139
- [Background] Asar S, Rahim F, Rahimi P, Acicbe O, Tontu F, Cukurova Z. Novel Oxygenation and Saturation Indices for Mortality Prediction in COVID-19 ARDS Patients: The Impact of Driving Pressure and Mechanical Power. J Intensive Care Med. 2024 Jun;39(6):595-608. doi: 10.1177/08850666231223498. Epub 2024 Jan 5. PMID 38179691